CLINICAL TRIAL: NCT03784807
Title: New Strategies for Diagnosis and Management of Biofilm Related Infections
Brief Title: New Strategies for Biofilm Related Infections
Acronym: Diafilm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Diafilm
Record Dates: First submitted 2018-12-06; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Prosthetic Joint Infection
Keywords: synovial fluid analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial strains
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infected: Patients with prosthetic joint or osteoarticular infection
  Interventions: Diagnostic Test: synovial calprotectin, confocal laser microscopy
- Not infected: Patients with implant failure not due to infection
  Interventions: Diagnostic Test: synovial calprotectin, confocal laser microscopy

INTERVENTIONS:
Diagnostic Test: synovial calprotectin, confocal laser microscopy — Calprotectin will be determined in synovial fluid of patients with septic and aseptic failure of their prosthesis. CLSM will be used to detect presence of microorganisms in synovial fluid. Susceptibility to antimicrobials of bacterial strains isolated from patients with prosthetic joint infections will be assessed using planktonic cells and biofilm associated bacteria

SUMMARY:
This study aims to develop new assays for synovial fluid analysis able to improve diagnosis of prosthetic joint infections. In particular, use of synovial calprotectin as marker of infection, confocal laser scanning microscopy (CLSM) analysis and methods to assess antimicrobial susceptibility will be evaluated in synovial fluids collected from patients with septic and aseptic failure of the prosthetic implant.

DETAILED DESCRIPTION:
Infection of prosthetic joints is a common complication that may occur any time after implantation. These infections require a prompt and accurate diagnosis to ensure an optimal surgical and medical management of infected patient. Despite acute infections occurring in the first weeks after surgery are easy to diagnose or when they are associated to bacteremia, diagnosis becomes challenging when infection develops for several months before diagnosis or it is caused by low virulent pathogens. Prosthetic joint infections and more widely osteo-articular infections represent the classic biofilm related infections. Biofilm is usually defined as a microbial community enveloped in a self-produced polymeric matrix. Biofilm production allows bacteria to strictly adhere to inert and biotic substrates, evade host defenses and resist to antibiotics by building a physical barrier to penetration of antimicrobials and favoring dissemination of determinants of resistance. Microbiological cultures contribute to diagnosis of infection, providing identification of the pathogen and, most importantly, definition of antibiotic susceptibility. Nonetheless, in about 15-20% of cases, culture fails to growth the pathogen. Diagnosis of prosthetic joint infection may occur either pre- or intra-operatively. In both cases analysis of synovial fluid is crucial, especially when performed before surgery when results from culture, leukocyte esterase, alpha defensin test, leukocyte count and differential may lead to define the most accurate strategy to approach patients with implant failure. However, culture of synovial fluid is characterized by a limited sensitivity in respect, for instance to culture of periprosthetic tissues or implant components. One of the causes of the lower sensitivity of synovial fluid culture might be the presence of the so called "biofilm like aggregates", agglomerates of microorganisms embedded in a matrix which has been hypothesized to act as a protective barrier. Leukocyte esterase test may give false positive results in samples strongly contaminated by blood or with metal on metal reaction, while the high costs for alpha defensin determination markedly limited its use. On the other hand, studies aiming to evaluate other synovial markers of infections like calprotectin are insufficient to support their use in routine diagnosis of prosthetic joint infection.

An alternative approach to diagnosis of these infections could be represented by use of confocal laser scanning microscopy (CLSM) which allows to detect microorganisms in synovial fluid and in tissues. This novel approach could also be used for a "real time" diagnosis during surgery while waiting for culture results.

Another issue in diagnosis of prosthetic joint infections is related to assessment of antimicrobial susceptibility. In fact, it is well known that biofilm embedded bacteria are more resistant to antibiotics than their planktonic counterpart. Since available methods for determination of antibiotic susceptibility are based on planktonic cells, it may be hypothesized that they underestimate the real antimicrobial concentration able to inhibit growth of bacteria embedded in a biofilm as occur during infection. Although several methods have been proposed to evaluate antimicrobial susceptibility pattern of biofilm microorganisms, none of them has been proposed for routinely use. However, in some cases when therapy fails to eradicate infection, evaluation of antibiotic susceptibility of biofilm embedded bacteria could provide important information to optimize antimicrobial therapy.

Therefore, diagnosis of biofilm related infections, particularly prosthetic ones is quite far from being optimized. In this sense, development of a panel able to shorten turn around time of microbiological analyses and to improve patient management could significantly ameliorate approach to patients, limiting worsening in patient's quality of life and reducing costs for health system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of implant failure or osteoarticular infections
* Collection of a sufficient amount of synovial fluid
* Informed Consent signed

Exclusion Criteria:

* Patients not fulfilling the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoarticular or prosthetic joint infection
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of analytical performance of calprotectin and CLSM for diagnosis of prosthetic joint infections | preoperative visit or during surgery
  Sensitivity, specificity, predictive values and diagnostic accuracy of calprotectin and CLSM will be calculated and compared to those of assays already used for diagnosis of prosthetic joint infections

SECONDARY OUTCOMES:
Improvement in antibiotic therapy applying data obtained from antibiotic susceptibility testing on biofilm | Afetr isolation of the pathogen, within 2 months
  Antimicrobial profiles obtained on biofilm bacteria will be compared with those obtained with traditional methods on planktonic cells

CONTACTS AND LOCATIONS:
Overall Officials: Elena De Vecchi, MSc, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary outcomes measures for all participants to the study will be made available
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available within 1 year from study conclusion
Access Criteria: Requests should be sent by e-mail to the Institution